CLINICAL TRIAL: NCT01789801
Title: A Randomized Study Evaluating the Role of Ultra-sound Guidance When Drawing Radial Arterial Blood Samples
Acronym: ECHO-PARDIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2012/RGG-01; 2012-A01525-38 (Other: ANSM)
Record Dates: First submitted 2013-02-09; First posted 2013-02-12 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-06

CONDITIONS: Radial Artery; Ultrasonography
MeSH Terms: interventions — LDL-Receptor Related Protein-Associated Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation only (Active Comparator): Patients randomized to this arm will have radial artery puncture via palpation of arteries.
  Intervention: RAP palpation only
  Interventions: Procedure: RAP palpation only
- Ultrasound guidance (Experimental): Patients randomized to this arm will have radial artery puncture with ultrasound guidance for artery localisation.
  Intervention: RAP with ultrasound guidance
  Interventions: Procedure: RAP with ultrasound guidance

INTERVENTIONS:
Procedure: RAP palpation only — Skin disinfection by local antiseptic. Identification of the radial artery by palpation. Insertion of the needle positioned at 70 ° with regard to the artery palpated. Check the rise of arterial blood in the syringe.
  Other Names: Radial artery puncture via palpation of arteries only
  Arms: Palpation only
Procedure: RAP with ultrasound guidance — Skin disinfection by local antiseptic. Application of sterile gel. Identification of the artery via ultrasound vascular probe. Center the artery at the center of the screen. Introduction of the syringe at 70 ° with respect to the probe, in center of visualized zone. Check the rise of arterial blood in the syringe.
  Other Names: radial artery puncture with ultrasound guidance.
  Arms: Ultrasound guidance

SUMMARY:
Previous studies have demonstrated that an experienced ultrasound operator is able to efficiently perform radial arterial puncture on patients where an initial operator failed to puncture arteries via simple palpation.

The objective of this study is to compare "difficult-to-puncture" patients randomized into two groups: one group where ultrasound is used to aid artery localisation, and one group where only palpation is used.

DETAILED DESCRIPTION:
test

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient's health status necessitates an arterial blood sample AND his/her radial arteries are deemed unpalpable OR two previous attempts at radial arterial puncture by a nurse resulted in failure

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or any kind of guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Arterial puncture is required on femoral, humeral or axillary arteries
* The patient is in cardiac arrest
* The patient has known circulatory problems, ischemia, local infection
* The patient has a severe bleeding or hemostasis disorder (hemophilia, hypoprothrombinemia, platelets <50,000)
* The patient is an upper limb amputee, or his/her arm is in a cast
* The patient has known allergies to methyl or propylbenzoate, propylene glycol or chlorexhidine gluconate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Only one attempt at arterial puncture was necessary (yes/no) | Day 0 - end of procedure

SECONDARY OUTCOMES:
Number of skin punctures | Day 0 - end of procedure
Length of time necessary for the procedure | Day 0 - end of procedure
Presence/absence of complications | Day 0 - end of procedure
  Presence/absence of complications including hematoma, nerve injury, vagal reaction, pseudo-aneurysm.
Patient satisfaction | Day 0 - end of procedure
  Patient satisfaction is evaluated using a visual analog scale.
Operator satisfaction | Day 0 - end of procedure
  Operator satisfaction is estimated using a visual analog scale.
Patient pain evaluation | Day 0 - end of procedure
  Patients are asked to evaluate the experienced pain level using a visual analog scale.
The number of catheters used | Day 0 - end of procedure
Was additional assistance necessary? yes/no | Day 0 - end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Romain Genre-Grandpierre, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Genre Grandpierre R, Bobbia X, Muller L, Markarian T, Occean BV, Pommet S, Roger C, Lefrant JY, de la Coussaye JE, Claret PG. Ultrasound guidance in difficult radial artery puncture for blood gas analysis: A prospective, randomized controlled trial. PLoS One. 2019 Mar 20;14(3):e0213683. doi: 10.1371/journal.pone.0213683. eCollection 2019. PMID 30893349
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140